CLINICAL TRIAL: NCT02609880
Title: Cognitive Behavioral Effects on Sleep, Pain, and Cytokines in Gynecologic Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: University of Miami (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB201600679-N; R01CA138808 (NIH); 287-2009 (Other: University of Florida)
Record Dates: First submitted 2015-11-09; First posted 2015-11-20 (Estimated); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Genital Neoplasms, Female; Insomnia; Pain; Adaptation, Psychological
Keywords: Psycho-Oncology; Psychoneuroimmunology; Cognitive Behavioral Therapy; Gynecologic Cancer; Insomnia; Pain; Distress; Cortisol; Cytokines
MeSH Terms: conditions — Genital Neoplasms, Female; Sleep Initiation and Maintenance Disorders; Pain | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Behavioral Therapy (Experimental): This group will receive Cognitive Behavioral Therapy to optimize sleep, pain, and mood in women with gynecologic cancers. The therapy will be provided on a one-on-one basis, for 2 hours once a week for six weeks by a trained therapist with a master's degree in Clinical Psychology.
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Psychoeducation (Placebo Comparator): This group will receive Psychoeducation which is aimed at providing information, resources, and non-specific support related to adapting well to cancer. The education will be provided on a one-on-one basis, for 2 hours once a week for six weeks by a trained therapist with a master's degree in Clinical Psychology.
  Interventions: Behavioral: Psychoeducation

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Cognitive Behavioral Therapy is used to optimize sleep, pain, and mood in women with gynecologic cancers and will be provided 2 hours once a week for six weeks.
  Arms: Cognitive Behavioral Therapy
Behavioral: Psychoeducation — Psychoeducation is used to provide information, resources, and non-specific support related to adapting well to cancer. Sessions will be provided 2 hours once a week for 6 weeks.
  Arms: Psychoeducation

SUMMARY:
Gynecologic cancers cause substantial morbidity and mortality among women. Developing, implementing, and disseminating interventions that reduce morbidity and mortality secondary to gynecologic cancers are a public health priority. In spite of this, there is a paucity of research examining the effects of psychosocial interventions on patient-centered and physiological outcomes in this population. To the extent that psychological factors may influence quality of life and tumor biology among women with gynecologic cancers, psychological interventions may represent an important adjunct to standard clinical care in this population. As such, this study will examine the effects of a psychosocial intervention on sleep, pain, mood, cortisol, and cytokines in women with gynecologic cancers.

DETAILED DESCRIPTION:
Gynecologic cancers cause substantial morbidity and mortality among women. Developing, implementing, and disseminating interventions that reduce morbidity and mortality secondary to gynecologic cancers are a public health priority. To the extent that psychological factors may influence quality of life and tumor biology among women with gynecologic cancers, psychological interventions may represent an important adjunct to standard clinical care in this population. Among individuals with cancer, there is emerging evidence that stressors and psychological responses to stressors activate central and peripheral stress systems, resulting in downstream effects on the tumor microenvironment, e.g. hypothalamic-pituitary-adrenal (HPA) axis dysregulation, inflammatory/growth factor upregulation that may favor tumorigenesis. Little is known about whether psychological interventions may modulate biobehavioral factors that may promote tumorigenesis among women with gynecologic cancer. This is a significant gap in the literature. Sleep quality, pain, and mood are three patient-centered outcomes that may represent important intervention targets for women with gynecologic cancers, as insomnia, pain, and negative mood states are (1) prevalent and (2) have been associated with HPA dysregulation and inflammatory/growth factor upregulation in this population in empirical research. This study will examine cognitive behavioral therapy (CBT) intervention effects on patient centered and physiological outcomes among women with gynecologic cancers undergoing adjuvant chemotherapy. Grounded within the Central Arousal Theory of Stress (CATS) and a biobehavioral model of tumor biology, the central hypothesis is that a CBT intervention targeting insomnia and pain will (a) improve nighttime sleep patterns, pain, and negative mood states, and (b) reduce cortisol levels, normalize daytime cortisol rhythm, and reduce proinflammatory/proangiogenic cytokine levels in women with gynecologic cancers. The multidisciplinary team will have research/clinical experience in psycho-oncology, psychoneuroimmunology (PNI), behavioral sleep medicine, pain, reproductive immunology, and gynecologic oncology. The research study is innovative in that it will (1) combine empirically-supported CBT techniques for insomnia and pain into a multicomponent intervention tailored for women with gynecologic cancers, and (2) examine CBT effects on central sensitization of pain among individuals with cancer using quantitative sensory testing (QST). The results of this research will be significant to public health initiatives, because although gynecologic cancers are among the leading causes of cancer-related death among women, there is a paucity of research examining the effects of psychosocial interventions on patient-centered and physiological outcomes in this population.

ELIGIBILITY:
Inclusion Criteria

* Women 18 and older scheduled and/ or have recently had a surgical resection, debulking, or cytoreduction for gynecologic malignancies for which adjuvant treatment or chemotherapy is the standard of care. Most of these cases are expected to be: (i) epithelial ovarian cancer, any stage, any grade, (ii) epithelial endometrial cancer, clear cell, papillary serous, or carcinosarcoma morphologies; any stage; any grade, (iii) epithelial endometrial cancer, endometrioid morphology; any stage any grade, (iv) fallopian tube cancer, any stage, any grade, (v) peritoneal cancer, any stage, any grade, or (vi) squamous cell carcinomas of the female genital tract (uterus, cervix, vulva, and vagina), any stage, any grade, in situ, or (vii) borderline ovarian tumors.
* Endorsement of any of the following sleep related complaints in the month prior to enrollment (at pre- or post-surgery): difficulty initiating sleep, difficulty maintaining sleep, waking up too early, or sleep that is chronically nonrestorative or poor in quality.
* During the two weeks of sleep evaluation at the post-surgical timepoint: sleep diary/clinical interview confirmed insomnia (e.g., sleep onset or awake time during the night > 30 minutes) at least 3 nights per week; or, sleep diary/clinical interview confirmed insomnia on 1 to 5 nights across the two weeks of evaluation plus Sleep Efficiency on Pittsburgh Sleep Quality Index at post-surgery < 85%.
* Presence of daytime dysfunction due to insomnia (mood, cognitive, social, or occupational impairment) at post-surgery.
* Able to read and understand English.
* Willing to undergo randomization.

Exclusion Criteria:

* Unable to provide informed consent.
* Current, severe, uncontrolled psychopathology that would make randomization to conditions unethical.
* Past or current diagnosis of Bipolar Disorder or seizure disorder that would prevent the safe implementation of sleep restriction techniques.
* Participation in Cognitive Behavioral Therapy or any nonpharmacological treatment for sleep outside of the current study.
* Sleep apnea or periodic limb movement disorder (PLMD).
* Physician estimated survival less than 6 months.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2009-07 (Actual); Primary Completion 2019-04-18 (Actual); Study Completion 2023-05-02 (Actual)

PRIMARY OUTCOMES:
Subjective Sleep Efficiency | Pre-surgery (T0, which is baseline), 6-8 weeks (T1, which is post-surgery and pre-intervention), 12-16 weeks (T2, which is post-intervention), and 18-24 weeks (T3, which is follow-up)
  Subjective Sleep Efficiency is assessed using daily Sleep Diaries.
  Analyses will examine intervention effects on changes in Sleep Efficiency from T1 to T2 and T1 to T3.
Subjective Sleep Quality | Pre-surgery (T0, which is baseline), 6-8 weeks (T1, which is post-surgery and pre-intervention), 12-16 weeks (T2, which is post-intervention), and 18-24 weeks (T3, which is follow-up)
  Subjective Sleep Quality is assessed using daily Sleep Diaries.
  Analyses will examine intervention effects on changes in Sleep Quality from T1 to T2 and T1 to T3.
Pain Quality and Intensity | Pre-surgery (T0, which is baseline), 6-8 weeks (T1, which is post-surgery and pre-intervention), 12-16 weeks (T2, which is post-intervention), and 18-24 weeks (T3, which is follow-up)
  Pain quality and intensity are assessed with the McGill Pain Questionnaire (MPQ) Total Score.
  Analyses will examine intervention effects on changes in pain severity from T1 to T2 and T1 to T3 while controlling for T0.
Pain Severity | Pre-surgery (T0, which is baseline), 6-8 weeks (T1, which is post-surgery and pre-intervention), 12-16 weeks (T2, which is post-intervention), and 18-24 weeks (T3, which is follow-up)
  Pain Severity is assessed using daily sleep Diaries.
  Analyses will examine intervention effects on changes in Pain Severity from T1 to T2 and T1 to T3.
Pain Interference | Pre-surgery (T0, which is baseline), 6-8 weeks (T1, which is post-surgery and pre-intervention), 12-16 weeks (T2, which is post-intervention), and 18-24 weeks (T3, which is follow-up)
  Pain Interference is assessed with the Pain Disability Index (PDI).
  Analyses will examine intervention effects on changes in Pain Disability from T1 to T2 and T1 to T3 while controlling for T0.
Serum Cortisol Concentrations | Pre-surgery (T0, which is baseline), 6-8 weeks (T1, which is post-surgery and pre-intervention), 12-16 weeks (T2, which is post-intervention), and 18-24 weeks (T3, which is follow-up)
  Serum Cortisol Concentrations are assessed with peripheral venous blood draw.
  Analyses will examine intervention effects on changes in Serum Cortisol Concentrations from T1 to T2 and T1 to T3 controlling for T0.
Diurnal Salivary Cortisol Rhythm | Pre-surgery (T0, which is baseline), 6-8 weeks (T1, which is post-surgery and pre-intervention), 12-16 weeks (T2, which is post-intervention), and 18-24 weeks (T3, which is follow-up)
  Diurnal Salivary Cortisol Rhythm is assessed with saliva sampling.
  Analyses will examine intervention effects on changes in Diurnal Salivary Cortisol Rhythm from T1 to T2 and T2 to T3 controlling for T0.
Serum Cytokine Concentrations | Pre-surgery (T0, which is baseline), 6-8 weeks (T1, which is post-surgery and pre-intervention), 12-16 weeks (T2, which is post-intervention), and 18-24 weeks (T3, which is follow-up)
  Cytokines are assessed by measuring serum concentrations of Interleukin (IL)-1, IL-6, IL-8, Tumor Necrosis Factor (TNF)-alpha, and Vascular Endothelial Growth Factor (VEGF).
  Analyses will examine intervention effects on changes in Cytokine Concentrations from T1 to T2 and T1 to T3 controlling for T0.

SECONDARY OUTCOMES:
Depressed Mood | Pre-surgery (T0, which is baseline), 6-8 weeks (T1, which is post-surgery and pre-intervention), 12-16 weeks (T2, which is post-intervention), and 18-24 weeks (T3, which is follow-up)
  Depressed Mood is assessed using the GRID-Hamilton Rating Scale for Depression (GRID-HAMD).
  Analyses will examine intervention effects on changes on GRID-HAMD scores from T1 to T2 and T1 to T3 controlling for T0.
Anxious Mood | Pre-surgery (T0, which is baseline), 6-8 weeks (T1, which is post-surgery and pre-intervention), 12-16 weeks (T2, which is post-intervention), and 18-24 weeks (T3, which is follow-up)
  Anxious mood is assessed via the State-Trait Anxiety Inventory (STAI).
  Analyses will examine intervention effects on changes on STAI State Anxiety scores from T1 to T2 and T1 to T3 controlling for T0.
A-Delta Nerve Fiber (First Pain) Response | Pre-surgery (T0, which is baseline), 6-8 weeks (T1, which is post-surgery and pre-intervention), 12-16 weeks (T2, which is post-intervention), and 18-24 weeks (T3, which is follow-up)
  This is assessed by measuring pain severity ratings in response to Graded Thermal Stimulation or RAMP and HOLD using Quantitative Sensory Testing.
  Analyses will examine intervention effects on changes in pain severity ratings from T1 to T2 and T1 to T3.
C Nerve Fiber (Second Pain) Response | Pre-surgery (T0, which is baseline), 6-8 weeks (T1, which is post-surgery and pre-intervention), 12-16 weeks (T2, which is post-intervention), and 18-24 weeks (T3, which is follow-up)
  This is assessed by measuring pain severity ratings in response to a Thermal Protocol for Temporal Summation or Wind-Up using Quantitative Sensory Testing
  Analyses will examine intervention effects on changes in pain severity ratings from T1 to T2 and T1 to T3.

CONTACTS AND LOCATIONS:
Overall Officials: Deidre B. Pereira, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Result] Padron A, McCrae CS, Robinson ME, Waxenberg LB, Antoni MH, Berry RB, Castagno J, Schultz G, Kacel EL, Ulfig C, Garey S, Patidar S, Sannes T, Trinastic L, Wong S, Pereira DB. Impacts of Cognitive Behavioral Therapy for Insomnia and Pain on Sleep in Women with Gynecologic Malignancies: A Randomized Controlled Trial. Behav Sleep Med. 2022 Jul-Aug;20(4):460-476. doi: 10.1080/15402002.2021.1932500. Epub 2021 Jun 14. PMID 34124972
- [Result] Hanvey GA, Padron A, Kacel EL, Cartagena G, Bacharz KC, McCrae CS, Robinson ME, Waxenberg LB, Antoni MH, Berry RB, Schultz GS, Castagno J, Pereira DB. Accrual and retention of diverse patients in psychosocial cancer clinical trials. J Clin Transl Sci. 2022 Apr 1;6(1):e45. doi: 10.1017/cts.2022.380. eCollection 2022. PMID 35651964
- [Derived] Cai Z, Tang Y, Liu C, Li H, Zhao G, Zhao Z, Zhang B. Cognitive behavioural therapy for insomnia in people with cancer. Cochrane Database Syst Rev. 2025 Oct 31;10(10):CD015176. doi: 10.1002/14651858.CD015176.pub2. PMID 41170811
- [Derived] Kacel EL, Kirsch JL, Sannes TS, Patidar S, Postupack R, Jensen S, Wong S, Garey S, Dodd S, Ulfig CM, McCrae CS, Robinson ME, Castagno J, Schultz GS, Pereira DB. Interleukin-6 and body mass index, tobacco use, and sleep in gynecologic cancers. Health Psychol. 2019 Oct;38(10):866-877. doi: 10.1037/hea0000775. Epub 2019 Aug 1. PMID 31368718
- [Derived] Kirsch JL, Robinson ME, McCrae CS, Kacel EL, Wong SS, Patidar S, Sannes TS, Garey S, Castagno JC, Pereira DB. Associations Among Sleep Latency, Subjective Pain, and Thermal Pain Sensitivity in Gynecologic Cancer. Pain Med. 2020 Jan 1;21(1):5-12. doi: 10.1093/pm/pny236. PMID 30481329